CLINICAL TRIAL: NCT06693310
Title: STOP-UC: De-escalation of Therapy in Patients With Ulcerative Colitis With Histological Remission
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB24-0008
Record Dates: First submitted 2024-11-07; First posted 2024-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC)
Keywords: histological remission; de-escalation of therapy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): continuation of current therapy
  Interventions: Other: continuation of current therapy
- de-escalation group (Active Comparator): de-escalation or discontinuation of therapy
  Interventions: Other: de-escalation or discontinuation of therapy

INTERVENTIONS:
Other: de-escalation or discontinuation of therapy — De-escalation of therapy, defined as a step-down from maintenance with advanced therapy (biologic or synthetic small molecule) to oral aminosalicylate-based therapy or complete discontinuation of therapy if they are allergic or intolerant to aminosalicylate-based therapy. If patients are receiving immunomodulator or oral aminosalicylate maintenance therapy, they will be de-escalated to complete discontinuation of therapy.
  Arms: de-escalation group
Other: continuation of current therapy — continuation of current maintenance medical therapy for ulcerative colitis
  Arms: Control group

SUMMARY:
The goal of this study is to better understand treatment strategies for people with ulcerative colitis (UC). Researchers will compare patients with UC in histologic remission (no evidence of inflammation or active disease on endoscopy and biopsies) who continue to take medical therapy to patients with UC who de-escalate (decrease or discontinue) medical therapy. Both treatment strategies are considered within regular medical practice. Researchers want to find out whether remission can be maintained after de-escalation of therapy.

Participants will be:

* either be randomly assigned to continue medical therapy or de-escalate medical therapy -OR- be assigned per the participant's preference
* clinically managed according to regular medical care
* asked to provide blood, stool (poop), and tissue samples for study purposes

DETAILED DESCRIPTION:
This is a prospective, partially-randomized, patient-preference clinical trial conducted at a tertiary academic center [University of Chicago Medicine Inflammatory Bowel Disease (IBD) Center]. Patients in clinical, biochemical, and endoscopic remission with biopsies showing histologic quiescence or normalization will be identified and approached after consultation with their IBD care team.

Subjects will be given a choice to either de-escalate their therapy (de-escalation group) or continue their current therapy (control group). This study design is to enhance the feasibility and real-world applicability. By permitting participants with strong preferences to choose their assigned strategy, we anticipate higher enrollment and retention among eligible subjects who might otherwise decline participation. Participants without a clear preference will be randomized 1:1 to de-escalation versus continuation, thereby preserving the integrity of comparative analyses. This approach enhances generalizability, respects patient autonomy, and mirrors clinical decision-making in routine clinical practice while maintaining methodological rigor.

After enrollment, participants will be monitored for 24 months. After the 24-month period, participants who remain in remission will continue 5 years of longitudinal data collection from routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting patients aged 18 to 75 years with an established diagnosis of ulcerative colitis (UC) for at least 3 years.
2. Patients in deep remission, defined by the absence of endoscopic and histologic signs of active inflammation (i.e. histological normalization or histological quiescence) in all biopsies obtained during colonoscopy, within the last 12 months.

   * If the most recent colonoscopy is within the last 3 years and demonstrates normalized/quiescent pathology findings (i.e., patient is in stable remission), the patient would not be expected to undergo yearly colonoscopies. Therefore, a persistent normalized calprotectin test will be accepted as sufficient to define deep remission with no change in therapy.
3. Patients in clinical, biochemical (fecal calprotectin <100), radiologic and endoscopic remission since the last colonoscopy.

Exclusion Criteria:

1. Any noted active inflammation [clinical, sonographic, biochemical, endoscopic (in any colonic segment)].
2. Patients with any changes in therapy after colonoscopy showing histological normalization or quiescence.
3. Corticosteroid use after colonoscopy showing histologic normalization or quiescence.
4. Patients with any noted history of primary sclerosing cholangitis or invisible or unresected high-grade dysplasia (suspected or confirmed).
5. Pregnancy or actively trying to conceive
6. Inability to follow the proposed sample collection and monitoring protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of individuals with sustained biochemical remission | Baseline, 12 months
  Biochemical remission defined as fecal calprotectin (FCP) level less than 150 and C-reactive protein (CRP) level less than the predetermined normal range according to the test manufacturer (typically less than 5.0mg/dL).
Number of individuals with sustained sonographic remission | Baseline, 12 months
  Sonographic remission defined as bowel wall thickness (BWT) less than 4 millimeters(mm) in rectum and BWT less than 3 mm in the remainder of the bowel; measured by intestinal ultrasound
Number of individuals with sustained clinical remission | Baseline, 12 months
  Clinical remission defined as Patient-Reported Outcome (PRO-2) score less than 1. The PRO-2 questionnaire measures patient-reported stool frequency and rectal bleeding in UC; scores range from 0-3, with higher scores indicating more severe symptoms.
Number of individuals with sustained endoscopic remission | Baseline, 12 months
  Endoscopic remission defined as Mayo endoscopic subscore equal to 0 or 1. The Mayo endoscopic subscore is a physician-reported measure of mucosal appearance at endoscopy. Scores range from 0-3, with higher scores indicating more disease activity.

SECONDARY OUTCOMES:
Proportion of individuals maintaining corticosteroid-free remission | 12 months
  Calculated by dividing the number of individuals maintaining remission without the need for corticosteroid medications by the total number of individuals in the study
Change in host metabolites in states of deep remission | Baseline, at the time points when deep remission is clinically confirmed (expected at scheduled assessments at 6, 12, 18, and 24 months)
  Measured by mass spectrometry, flow cytometry, enzyme-linked immunosorbent assay (ELISA)-based assays and/or real-time polymerase chain reaction (RT-PCR)-based assays
Change in microbial metabolites in states of deep remission | Baseline, at the time points when deep remission is clinically confirmed (expected at scheduled assessments at 6, 12, 18, and 24 months)
  Quantitative measurement of host metabolites using mass spectrometry, flow cytometry, enzyme-linked immunosorbent assays (ELISA), and/or real-time polymerase chain reaction (RT-PCR)-based assays to characterize biochemical changes associated with deep remission
Change in host metabolites in states of disease relapse | Baseline, at the time points when deep remission is clinically confirmed (expected at scheduled assessments at 6, 12, 18, and 24 months)
  Measured by mass spectrometry, flow cytometry, ELISA-based assays and/or RT-PCR-based assays
Change in microbial metabolites in states of disease relapse | Baseline, at the time points when deep remission is clinically confirmed (expected at scheduled assessments at 6, 12, 18, and 24 months)
  Measured by mass spectrometry, flow cytometry, ELISA-based assays and/or RT-PCR-based assays
Change in microbial composition in states of deep remission | Baseline, at the time points when deep remission is clinically confirmed (expected at scheduled assessments at 6, 12, 18, and 24 months)
  Measured by mass spectrometry and RT-PCR-based assays
Change in microbial abundance in states of deep remission | Baseline, at the time points when deep remission is clinically confirmed (expected at scheduled assessments at 6, 12, 18, and 24 months)
  Measured by RT-PCR-based assays
Change in microbial composition in states of disease relapse | Baseline, at the time points when deep remission is clinically confirmed (expected at scheduled assessments at 6, 12, 18, and 24 months)
  Measured by RT-PCR-based assays
Change in microbial abundance in states of disease relapse | Baseline, at the time points when deep remission is clinically confirmed (expected at scheduled assessments at 6, 12, 18, and 24 months)
  Measured by RT-PCR-based assays
Number of individuals with long-term remission | Month 24
  Remission defined as an individual with all of the following:
  1. Clinical remission: PRO-2 less than 1
  2. Biochemical remission: FCP less than 150, CRP less than 1.0 mg/dL
  3. Sonographic remission: BWT ultrasound assessment less than 4mm in Rectum; less than 3mm in remainder of Bowel
  4. Endoscopic remission: Mayo Endoscopic Subscore equals 0 or 1

CONTACTS AND LOCATIONS:
Overall Officials: David T Rubin, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States